CLINICAL TRIAL: NCT00457522
Title: Phone Intervention to Increase Safety in Abused Women: Pilot
Brief Title: Telephone Intervention to Increase Safety in Abused Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00001492; P30NR008995 (NIH)
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Intimate Partner Violence
Keywords: intimate partner violence; depression; PTSD; fatigue
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Fatigue | interventions — Nurses

INTERVENTIONS:
Behavioral: Nurse/community health worker telephone intervention

SUMMARY:
Although abuse by an intimate partner is very common and has serious negative effects on women's health, few studies have been done to test ways to increase safety for women in abusive relationships. This study will test a telephone intervention for women who report physical, emotional, and/or sexual abuse within the past 12 months, to see if

* women use more safety behaviors and access more community resources
* chronic pain, fatigue, depressive, and post-traumatic stress disorder (PTSD) symptoms affect a women's ability to use safety behaviors and access community resources.

DETAILED DESCRIPTION:
Women who experience intimate partner violence (IPV) are at increased risk for serious long term negative health sequelae, injury, and death. Compared to non-abused women, intimately abused women suffer significantly greater prevalence of depression and post-traumatic stress disorder (PTSD), as well as a host of nonspecific physical symptoms including chronic pain and fatigue (Campbell, 2002; Golding, 1999; Asmundson, Coons, Taylor, & Katz, 2002; Ehlert, Gaab, & Heinrichs, 2001; Green, Baker, Sato, Washington, & Smith, 2003; Woods, 2004). These increased negative health problems contribute to a greater prevalence of IPV among primary care patients, with current (past year) IPV rates of 15 - 28%, compared to 1.5% to 3% in epidemiologic surveys (Bauer, Rodruguez, Perez-Stable, 2000; Coker, et al., 2000; Collins, et al.,1998; Kramer, Lorenzon, Mueller, 2004; Richardson, et al., 2002; Tjaden & Thoennes, 2000). In spite of this high prevalence and serious negative health sequelae, a recent review of interventions for IPV concluded that there is a serious lack of evidence-based approaches in the primary care setting. No studies were identified that examined the effect of physical and mental health symptoms on the ability to access resources or to increase safety promoting behaviors. This intervention pilot study will speak to this gap in the research. Utilizing a randomized controlled clinical trial design, we will follow women who screen positive for current (past year) IPV at a primary care clinic in Baltimore, MD. Women in the control group will receive usual care consisting of a list of community resources for IPV. Women in the a nurse-managed/community health worker intervention group will receive usual care augmented by an individualized counseling session followed by a series of 6 telephone calls over 10 weeks. A woman's stage of readiness for change as well as symptoms of pain, fatigue, depression, and PTSD will be evaluated as barriers to resource access and safety behavior initiation.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 years of age or older
* speaks English
* reports physical, emotional, and/or sexual abuse by an intimate partner within past 12 months

Exclusion Criteria:

* non-English speaking
* currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of safety promotion behaviors at initiation and completion of intervention
Number of community resources accessed at initiation and completion of intervention

SECONDARY OUTCOMES:
Stage of readiness for change at initiaion and completion of intervention
Severity of pain, fatigue, depressive and PTSD symptoms at initiation and completion of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Woods, PhD, CNM, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- The Shepherd's Clinic, Baltimore, Maryland, United States